CLINICAL TRIAL: NCT00398476
Title: A Patient Preference Evaluation Study of Fluticasone Furoate Nasal Spray and Fluticasone Propionate Aqueous Nasal Spray in Subject With Allergic Rhinitis
Brief Title: Fluticasone Nasal Spray Patient Preference Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Purpose: Treatment
Other Study IDs: FFU108556
Record Dates: First submitted 2006-11-09; First posted 2006-11-10 (Estimated); Results first posted 2018-01-29 (Actual); Last update posted 2018-03-01 (Actual); Status verified 2017-06

CONDITIONS: Rhinitis, Allergic, Perennial
Keywords: taste; questionnaire; preference; attributes; odor; after taste; scent
MeSH Terms: conditions — Rhinitis, Allergic, Perennial | interventions — Fluticasone; fluticasone furoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- fluticasone propionate (FP) (Active Comparator): 200 micrograms (mcg); an aqueous suspension of microfine FP
  Interventions: Drug: fluticasone propionate (FP)
- fluticasone furoate (FF) (Active Comparator): 110 mcg; an aqueous suspension containing 0.05% w/w of micronized FF
  Interventions: Drug: fluticasone furoate (FF)

INTERVENTIONS:
Drug: fluticasone propionate (FP) — 200 micrograms (mcg); an aqueous suspension of microfine FP
  Arms: fluticasone propionate (FP)
Drug: fluticasone furoate (FF) — 110 mcg; an aqueous suspension containing 0.05% w/w of micronized FF
  Other Names: fluticasone furoate; fluticasone propionate
  Arms: fluticasone furoate (FF)

SUMMARY:
The objectives of this study are to evaluate and compare patient preference for FF (Fluticasone Furoate) and FP (Fluticasone Propionate Aqueous)nasal sprays in the treatment of allergic rhinitis following single-dose administration.

ELIGIBILITY:
Inclusion Criteria:

* allergic rhinitis
* literate

Exclusion Criteria:

* clinical significant uncontrolled disease
* Use of intranasal corticosteroids (<4 weeks of FP [branded or generic],<4 week exposure to FF, <4 weeks use of other INS)
* Use of intranasal medications <1 week
* Use of meds that significantly inhibit CYP4503A4
* Use of perfume or oral rinse on study day
* Allergy/intolerance to INS, antihistamines, or excipients
* Positive pregnancy test or female who is breastfeeding
* Affiliation with investigational site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2006-12-01 (Actual); Primary Completion 2006-12-04 (Actual); Study Completion 2006-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (14):
- United States (14):
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Lakewood, Colorado
  - GSK Investigational Site, Lawrenceville, Georgia
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Ypsilanti, Michigan
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Rolla, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Brick, New Jersey
  - GSK Investigational Site, Skillman, New Jersey
  - GSK Investigational Site, El Paso, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 127 male or eligible female participants with a diagnosis of allergic rhinitis were enrolled in the study. This study was conducted at 12 investigator sites in the United States. Study duration was '01 December 2006 - 04 December 2006'. Participants included in PP population were 121.
Groups:
- FF 110 µg /FP 200 µg: In this sequence, participants received a single-dose treatment fluticasone furoate (FF) 110 micrograms (µg) in period 1 and fluticasone propionate (FP) 200 µg in period 2 (2 sprays per nostril - 4 sprays in total) for 30 minutes. Each spray of the suspension was containing approximately 27.5 µg of FF and each actuation delivered 50 µg of FP in 100 milligram (mg) of formulation through the nasal adapter. There was a washout period of 20 minutes in between the 2 periods.
- FP 200 µg /FF 110 µg: In this sequence, participants received a single-dose treatment FP 200 µg in period 1 and FF 110 µg in period 2 (2 sprays per nostril - 4 sprays in total) for 30 minutes. Each spray of the suspension was containing approximately 27.5 µg of FF and Each actuation delivered 50 µg of FP in 100 mg of formulation through the nasal adapter. There was a washout period of 20 minutes in between the 2 periods.
Period: Treatment Period 1
Arm/Group | FF 110 µg /FP 200 µg | FP 200 µg /FF 110 µg
Started | 63 | 64
Completed | 63 | 64
Not Completed | 0 | 0
Period: Washout Period (20 Minutes)
Arm/Group | FF 110 µg /FP 200 µg | FP 200 µg /FF 110 µg
Started | 63 | 64
Completed | 63 | 64
Not Completed | 0 | 0
Period: Treatment Period 2
Arm/Group | FF 110 µg /FP 200 µg | FP 200 µg /FF 110 µg
Started | 63 | 64
Completed | 63 | 64
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study Arm: Eligible participants were randomized (1:1) to receive a single-dose treatment (2 sprays per nostril - 4 sprays in total). Sequence of either FP 200 µg/FF 110 µg or FF 110 µg/FP 200 µgin a crossover manner. Prior to receiving the first treatment sequence, participants underwent a washout procedure, which consisted of cleaning the mouth by eating one unsalted followed by several swallows of room temperature water and sniffing a swatch of wool. Participants then received the first treatment in their randomization sequence (FF or FP, 2 sprays per nostril). Thirty minutes after the first treatment and prior to initialization of second washout period, Participants received the second treatment in their randomization sequence (FF or FP, 2 sprays per nostril). Participants completed two questionnaires, an immediate attributes questionnaire (administered immediately after dosing) followed by a delayed attributes questionnaire (administered 2 minutes after dosing).
Arm/Group | Overall Study Arm
Number analyzed (Participants) | 127
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.7 (14.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82
  Male | 45
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Intent to treat population comprised of all participants who were randomized to treatment with study drug. Where n was 126.
  Participants
    Race: number analyzed (Participants) | 126
    Race: African American/African Heritage | 20
    Race: Asian - East Asian Heritage | 1
    Race: Asian - South East Asian Heritage | 1
    Race: Native Hawaiian or other Pacific Islander | 1
    Race: White - Arabic/North African Heritage | 1
    Race: White - White/Caucasian/European Heritage | 100
    Race: Mixed Race | 2

OUTCOME MEASURES:

1. Primary Outcome: Overall Participants Preference for Nasal Spray Based on Selected Product Attributes at the End of Crossover Dosing
Description: An overall preference questionnaire (OPQ) was used to evaluate participant's preference for nasal spray therapy for the given treatments. OPQ allows the responder three options, based on products attributes, i.e. preference for product 1 (FF 110 µg); preference for product 2 (FP 200 µg) and no preference. Three participant-related questionnaires were completed during the course of the study, including two attributes questionnaires : Immediate attributes questionnaire (IAQ) and delayed attributes questionnaire (DAQ). An OPQ was completed upon completion of the crossover dosing.
Time Frame: Day 1
Population: Per Protocol population comprised of all participants who completed both treatment periods. Only those participants available at the indicated time points were analyzed.
Measure: Number; unit: Participants
Groups:
- Overall Study Arm: Eligible participants were randomized (1:1) to receive a single-dose treatment (2 sprays per nostril - 4 sprays in total). Sequence of either FP 200 µg /FF 110 µg or FF 110 µg /FP 200 µg in a crossover manner. Prior to receiving the first treatment sequence, participants underwent a washout procedure, which consisted of cleaning the mouth by eating one unsalted followed by several swallows of room temperature water and sniffing a swatch of wool. Participants then received the first treatment in their randomization sequence (FF or FP, 2 sprays per nostril). Thirty minutes after the first treatment and prior to initialization of second washout period, Participants received the second treatment in their randomization sequence (FF or FP, 2 sprays per nostril). Participants completed two questionnaires, an immediate attributes questionnaire (administered immediately after dosing) followed by a delayed attributes questionnaire (administered 2 minutes after dosing).
Arm/Group | Overall Study Arm
Number analyzed (Participants) | 120
Participants
  Overall, FF 110 µg | 72
  Overall, FP 200 µg | 39
  Overall, No preference | 9
  Scent/odor, FF 110 µg | 77
  Scent/odor, FP 200 µg | 35
  Scent/odor, No preference | 8
  Immediate taste, FF 110 µg | 56
  Immediate taste, FP 200 µg | 25
  Immediate taste, No preference | 39
  After-taste, FF 110 µg | 53
  After-taste, FP 200 µg | 26
  After-taste, No preference | 41
  Less drip down throat, FF 110 µg | 52
  Less drip down throat, FP 200 µg | 32
  Less drip down throat, No preference | 36
  Less run out nose, FF 110 µg | 59
  Less run out nose, FP 200 µg | 23
  Less run out nose, No preference | 38
  More soothing, FF 110 µg | 45
  More soothing, FP 200 µg | 38
  More soothing, No preference | 37
  Less irritating, FF 110 µg | 41
  Less irritating, FP 200 µg | 26
  Less irritating, No preference | 53
  Urge to sneeze, FF 110 µg | 25
  Urge to sneeze, FP 200 µg | 21
  Urge to sneeze, No preference | 74
Statistical Analysis 1: Comparison: Overall Study Arm; Analysis for overall product preference; Test type: Other; p = 0.003, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Overall Study Arm; Analysis for Scent/odor; Test type: Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Overall Study Arm; Analysis for Immediate taste; Test type: Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Overall Study Arm; Analysis for After-taste; Test type: Other; p = 0.002, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Overall Study Arm; Analysis for Less drip down throat; Test type: Other; p = 0.037, Cochran-Mantel-Haenszel
Statistical Analysis 6: Comparison: Overall Study Arm; Analysis for Less run out nose; Test type: Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 7: Comparison: Overall Study Arm; Analysis for More soothing; Test type: Other; p = 0.408, Cochran-Mantel-Haenszel
Statistical Analysis 8: Comparison: Overall Study Arm; Analysis for Less irritating; Test type: Other; p = 0.070, Cochran-Mantel-Haenszel
Statistical Analysis 9: Comparison: Overall Study Arm; Analysis for Urge to sneeze; Test type: Other; p = 0.587, Cochran-Mantel-Haenszel

2. Secondary Outcome: Number of Participants With Preference for Scent/Odor in IAQ and DAQ
Description: Participant preference for scent/odor at the end of crossover dosing with FF 110 µg and FP 200 µg was evaluated using IAQ and DAQ having question: Did product have a scent/odor?. Participants specified their responses on a 6-point scale: 0: none; 1: very mild; 2: mild; 3: neither mild nor strong; 4: slightly strong; 5; moderately strong; 6: very strong. Higher score indicated strong odor.
Time Frame: Day 1
Population: Per Protocol population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Participants
Groups:
- FF 110 µg: Participants were randomized to receive a single dose of FF 110 µg nasal spray (2 sprays per nostril - 4 sprays in total) for 30 minutes in treatment period 1 and 2. Each spray of the suspension was containing approximately 27.5 µg of FF. 2 attributes questionnaires (immediate and delayed) and an overall preference questionnaire were completed by participants during the course of the study.
- FP 200 µg: Participants were randomized to receive a single dose of FP 200 µg nasal spray (2 sprays per nostril - 4 sprays in total) for 30 minutes in treatment period 1 and 2. Each actuation delivered 50 µg of FP in 100 mg of formulation through the nasal adapter 2 attributes questionnaires (immediate and delayed) and an overall preference questionnaire were completed by participants during the course of the study.
Arm/Group | FF 110 µg | FP 200 µg
Number analyzed (Participants) | 121 | 121
Participants
  IAQ, None: number analyzed (Participants) | 121 | 120
  IAQ, None | 62 | 12
  DAQ, None | 71 | 16
  IAQ, Very mild: number analyzed (Participants) | 121 | 120
  IAQ, Very mild | 27 | 22
  DAQ, Very mild | 21 | 39
  IAQ, Mild: number analyzed (Participants) | 121 | 120
  IAQ, Mild | 19 | 35
  DAQ, Mild | 16 | 29
  IAQ, Neither mild nor strong: number analyzed (Participants) | 121 | 120
  IAQ, Neither mild nor strong | 2 | 7
  DAQ, Neither mild nor strong | 4 | 4
  IAQ, Slightly strong: number analyzed (Participants) | 121 | 120
  IAQ, Slightly strong | 6 | 20
  DAQ, Slightly strong | 6 | 20
  IAQ, Moderately strong: number analyzed (Participants) | 121 | 120
  IAQ, Moderately strong | 4 | 19
  DAQ, Moderately strong | 2 | 10
  IAQ, Very strong: number analyzed (Participants) | 121 | 120
  IAQ, Very strong | 1 | 5
  DAQ, Very strong | 1 | 3
Statistical Analysis 1: Comparison: FF 110 µg vs FP 200 µg; Comparison of FF 110 µg and FP 200 µg for IAQ items; Test type: Equivalence — Assuming that 65% of participants indicate an overall preference for FF over FP, then a sample size of 125 participants will provide 93% power to show that difference in proportions (i.e., 65% favoring FF vs 35% favoring FP); p < 0.001, Cochran-Mantel-Haenszel; Median Difference (Final Values) = -2.0
Statistical Analysis 2: Comparison: FF 110 µg vs FP 200 µg; Comparison of FF 110 µg and FP 200 µg for DAQ items; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; Median Difference (Final Values) = -1.0

3. Secondary Outcome: Number of Participants With Preference for Satisfaction With Scent/Odor in IAQ
Description: Participant preference for Satisfaction scent/odor at the end of crossover dosing with FF 110 µg and FP 200 µg was evaluated using IAQ having question: How satisfied with scent/odor?. Participants specified their responses on a 6-point scale: 0: very satisfied; 1: moderately satisfied; 2: somewhat satisfied; 3: neither satisfied nor dissatisfied; 4: somewhat dissatisfied; 5; moderately dissatisfied; 6: very dissatisfied.
Time Frame: Day 1
Population: Per protocol population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | FF 110 µg | FP 200 µg
Number analyzed (Participants) | 121 | 121
Participants
  IAQ, Very satisfied: number analyzed (Participants) | 61 | 109
  IAQ, Very satisfied | 11 | 16
  IAQ, Moderately satisfied: number analyzed (Participants) | 61 | 109
  IAQ, Moderately satisfied | 12 | 20
  IAQ, Somewhat satisfied: number analyzed (Participants) | 61 | 109
  IAQ, Somewhat satisfied | 13 | 25
  IAQ, Neither satisfied nor dissatisfied: number analyzed (Participants) | 61 | 109
  IAQ, Neither satisfied nor dissatisfied | 16 | 17
  IAQ, Somewhat dissatisfied: number analyzed (Participants) | 61 | 109
  IAQ, Somewhat dissatisfied | 6 | 23
  IAQ, Moderately dissatisfied: number analyzed (Participants) | 61 | 109
  IAQ, Moderately dissatisfied | 1 | 5
  IAQ, Very dissatisfied: number analyzed (Participants) | 61 | 109
  IAQ, Very dissatisfied | 2 | 3
Statistical Analysis 1: Comparison: FF 110 µg vs FP 200 µg; Comparison of FF 110 µg and FP 200 µg in IAQ; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.255, Cochran-Mantel-Haenszel; Median Difference (Net) = 0.0

4. Secondary Outcome: Number of Participants With Preference for Satisfaction With Scent/Odor in DAQ
Description: Participant preference for Satisfaction scent/odor at the end of crossover dosing with FF 110 µg and FP 200 µg was evaluated using IAQ and DAQ having question: How satisfied with scent/odor?. Participants specified their responses on a 6-point scale: 0: very satisfied; 1: moderately satisfied; 2: somewhat satisfied; 3: neither satisfied nor dissatisfied; 4: somewhat dissatisfied; 5; moderately dissatisfied; 6: very dissatisfied.
Time Frame: Day 1
Population: Per protocol population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | FF 110 µg | FP 200 µg
Number analyzed (Participants) | 53 | 106
Participants
  DAQ, Very satisfied | 14 | 19
  DAQ, Moderately satisfied | 11 | 21
  DAQ, Somewhat satisfied | 12 | 20
  DAQ, Neither satisfied nor dissatisfied | 10 | 22
  DAQ, Somewhat dissatisfied | 5 | 16
  DAQ, Moderately dissatisfied | 0 | 6
  DAQ, Very dissatisfied | 1 | 2
Statistical Analysis 1: Comparison: FF 110 µg vs FP 200 µg; Comparison of FF 110 µg and FP 200 µg for all DAQ items; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.056, Cochran-Mantel-Haenszel; Median Difference (Net) = 0.0

5. Secondary Outcome: Number of Participants Who Satisfied Not to Have Scent/Odor in IAQ
Description: Participant preference for participants who satisfied not to have scent/odor at the end of crossover dosing with FF 110 µg and FP 200 µg was evaluated using IAQ having question: How satisfied not to have scent/odor?. Participants specified their responses on a 6-point scale: 0: very satisfied; 1: moderately satisfied; 2: somewhat satisfied; 3: neither satisfied nor dissatisfied; 4: somewhat dissatisfied; 5; moderately dissatisfied; 6: very dissatisfied.
Time Frame: Day 1
Population: Per protocol population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | FF 110 µg | FP 200 µg
Number analyzed (Participants) | 121 | 121
Participants
  IAQ, Very satisfied: number analyzed (Participants) | 63 | 14
  IAQ, Very satisfied | 46 | 10
  IAQ, Moderately satisfied: number analyzed (Participants) | 63 | 14
  IAQ, Moderately satisfied | 7 | 2
  IAQ, Somewhat satisfied: number analyzed (Participants) | 63 | 14
  IAQ, Somewhat satisfied | 1 | 0
  IAQ, Neither satisfied nor dissatisfied: number analyzed (Participants) | 63 | 14
  IAQ, Neither satisfied nor dissatisfied | 6 | 1
  IAQ, Somewhat dissatisfied: number analyzed (Participants) | 63 | 14
  IAQ, Somewhat dissatisfied | 2 | 0
  IAQ, Moderately dissatisfied: number analyzed (Participants) | 63 | 14
  IAQ, Moderately dissatisfied | 0 | 0
  IAQ, Very dissatisfied: number analyzed (Participants) | 63 | 14
  IAQ, Very dissatisfied | 1 | 1
Statistical Analysis 1: Comparison: FF 110 µg vs FP 200 µg; Comparison of FF 110 µg and FP 200 µg for IAQ Irtems; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.845, Cochran-Mantel-Haenszel; Median Difference (Net) = 0.0

6. Secondary Outcome: Number of Participants Who Satisfied Not to Have Scent/Odor in DAQ
Description: Participant preference for participants who satisfied not to have scent/odor at the end of crossover dosing with FF 110 µg and FP 200 µg was evaluated using IAQ and DAQ having question: How satisfied not to have scent/odor?. Participants specified their responses on a 6-point scale: 0: very satisfied; 1: moderately satisfied; 2: somewhat satisfied; 3: neither satisfied nor dissatisfied; 4: somewhat dissatisfied; 5; moderately dissatisfied; 6: very dissatisfied.
Time Frame: Day 1
Population: Per protocol population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | FF 110 µg | FP 200 µg
Number analyzed (Participants) | 74 | 16
Participants
  DAQ, Very satisfied | 56 | 14
  DAQ, Moderately satisfied | 2 | 1
  DAQ, Somewhat satisfied | 4 | 0
  DAQ, Neither satisfied nor dissatisfied | 8 | 1
  DAQ, Somewhat dissatisfied | 3 | 0
  DAQ, Moderately dissatisfied | 0 | 0
  DAQ, Very dissatisfied | 1 | 0
Statistical Analysis 1: Comparison: FF 110 µg vs FP 200 µg; Comparison of FF 110 µg and FP 200 µg for DAQ Items; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.871, Cochran-Mantel-Haenszel; Median Difference (Net) = 0.0

7. Secondary Outcome: Number of Participants Reported Product Have an Immediate Taste in IAQ
Description: Participant preference for an immediate taste at the end of crossover dosing with FF 110 µg and FP 200 µg was evaluated using IAQ having question: Did product have an immediate taste?. Participants specified their responses on a on a 6-point scale: 0: no; 1: very mild; 2: mild; 3: neither mild nor strong; 4: slightly strong; 5; moderately strong; 6: very strong.
Time Frame: Day 1
Population: Per protocol population. Only those participants available at the indicated time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | FF 110 µg | FP 200 µg
Number analyzed (Participants) | 121 | 121
Participants
  No taste | 98 | 69
  Very mild taste | 10 | 25
  Mild taste | 7 | 13
  Neither mild nor strong taste | 2 | 6
  Slightly strong taste | 3 | 6
  Moderately strong taste | 1 | 2
  Very strong taste | 0 | 0
Statistical Analysis 1: Comparison: FF 110 µg vs FP 200 µg; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; Median Difference (Net) = 0.0

8. Secondary Outcome: Number of Participants Satisfied With an Immediate Taste in IAQ
Description: Participant preference for satisfaction with an immediate taste at the end of crossover dosing with FF 110 µg and FP 200 µg was evaluated using IAQ having question: How satisfied with immediate taste?. Participants specified their responses on a 6-point scale: 0: very satisfied; 1: moderately satisfied; 2: somewhat satisfied; 3: neither satisfied nor dissatisfied; 4: somewhat dissatisfied; 5; moderately dissatisfied; 6: very dissatisfied.
Time Frame: Day 1
Population: Per protocol population. Only those participants available at the indicated time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | FF 110 µg | FP 200 µg
Number analyzed (Participants) | 33 | 54
Participants
  Very satisfied | 6 | 12
  Moderately satisfied | 7 | 9
  Somewhat satisfied | 6 | 9
  Neither satisfied nor dissatisfied | 9 | 15
  Somewhat dissatisfied | 3 | 6
  Moderately dissatisfied | 1 | 3
  Very dissatisfied | 1 | 0
Statistical Analysis 1: Comparison: FF 110 µg vs FP 200 µg; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.592, Cochran-Mantel-Haenszel; Median Difference (Net) = 0.0

9. Secondary Outcome: Number of Participants Reported Product Have an After Taste in DAQ
Description: Participant response for an after taste at the end of crossover dosing with FF 110 µg and FP 200 µg was evaluated using DAQ having question: Did product have an aftertaste?. Participants specified their responses on a 6-point scale: 0: No aftertaste; 1: Very mild; 2: Mild; 3: Neither mild nor strong; 4: Slightly strong; 5: Moderately strong; 6: Very strong.
Time Frame: Day 1
Population: Per protocol population. Only those participants available at the indicated time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | FF 110 µg | FP 200 µg
Number analyzed (Participants) | 121 | 121
Participants
  No aftertaste | 90 | 66
  Very mild aftertaste | 22 | 33
  Mild aftertaste | 7 | 10
  Neither mild nor strong aftertaste | 0 | 3
  Slightly strong aftertaste | 2 | 6
  Moderately strong aftertaste | 0 | 3
  Very strong aftertaste | 0 | 0
Statistical Analysis 1: Comparison: FF 110 µg vs FP 200 µg; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; Median Difference (Net) = 0.0

10. Secondary Outcome: Number of Participants Satisfied With an After Taste in DAQ
Description: Participant response for satisfaction with an after taste at the end of crossover dosing with FF 110 µg and FP 200 µg was evaluated using DAQ having question: How satisfied with aftertaste? Participants specified their responses on a 6-point scale: 0: Very satisfied; 1: Moderately satisfied; 2: Somewhat satisfied; 3: Neither satisfied nor dissatisfied; 4: Somewhat dissatisfied; 5: Moderately dissatisfied; 6: Very dissatisfied.
Time Frame: Day 1
Population: Per protocol population. Only those participants available at the indicated time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | FF 110 µg | FP 200 µg
Number analyzed (Participants) | 34 | 54
Participants
  Very satisfied | 7 | 12
  Moderately satisfied | 8 | 9
  Somewhat satisfied | 3 | 7
  Neither satisfied nor dissatisfied | 11 | 15
  Somewhat dissatisfied | 3 | 9
  Moderately dissatisfied | 2 | 2
  Very dissatisfied | 0 | 0
Statistical Analysis 1: Comparison: FF 110 µg vs FP 200 µg; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.434, Cochran-Mantel-Haenszel; Median Difference (Net) = 0.0

11. Secondary Outcome: Number of Participants Reported Medicine Run Down Throat in IAQ and DAQ
Description: Participant response regarding did the medicine run down throat at the end of crossover dosing with FF 110 µg and FP 200 µg was evaluated using IAQ and DAQ having question: Did medicine run down throat? Participants specified their responses on a 6-point scale: 0: None; 1: Very slightly; 2: Slightly; 3: Neither slightly nor moderately; 4: Moderately; 5: Markedly; 6: Very markedly.
Time Frame: Day 1
Population: Per protocol population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | FF 110 µg | FP 200 µg
Number analyzed (Participants) | 121 | 121
Participants
  IAQ, None | 74 | 69
  DAQ, None: number analyzed (Participants) | 121 | 120
  DAQ, None | 64 | 55
  IAQ, Very slightly | 28 | 29
  DAQ, Very slightly: number analyzed (Participants) | 121 | 120
  DAQ, Very slightly | 36 | 37
  IAQ, Slightly | 11 | 15
  DAQ, Slightly: number analyzed (Participants) | 121 | 120
  DAQ, Slightly | 12 | 17
  IAQ, Neither slightly nor moderately | 3 | 5
  DAQ, Neither slightly nor moderately: number analyzed (Participants) | 121 | 120
  DAQ, Neither slightly nor moderately | 1 | 3
  IAQ, Moderately | 3 | 3
  DAQ, Moderately: number analyzed (Participants) | 121 | 120
  DAQ, Moderately | 5 | 6
  IAQ, Markedly | 1 | 0
  DAQ, Markedly: number analyzed (Participants) | 121 | 120
  DAQ, Markedly | 3 | 1
  IAQ, Very markedly | 1 | 0
  DAQ, Very markedly: number analyzed (Participants) | 121 | 120
  DAQ, Very markedly | 0 | 1
Statistical Analysis 1: Comparison: FF 110 µg vs FP 200 µg; This analysis is for IAQ; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.797, Cochran-Mantel-Haenszel; Median Difference (Net) = 0.0
Statistical Analysis 2: Comparison: FF 110 µg vs FP 200 µg; This analysis is for DAQ; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.296, Cochran-Mantel-Haenszel; Median Difference (Net) = 0.0

12. Secondary Outcome: Number of Participants Reported Medicine Run Out of Nose in IAQ and DAQ
Description: Participant response regarding did the medicine run out of nose at the end of crossover dosing with FF 110 µg and FP 200 µg was evaluated using IAQ and DAQ having question: Did medicine run out of nose? Participants specified their responses on a 6-point scale: 0: none; 1: very slightly; 2: slightly; 3: neither slightly nor moderately; 4: moderately; 5; markedly; 6: very markedly.
Time Frame: Day 1
Population: Per protocol population. Only those participants available at the indicated time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | FF 110 µg | FP 200 µg
Number analyzed (Participants) | 121 | 121
Participants
  IAQ, None | 61 | 38
  DAQ, None | 63 | 46
  IAQ, Very slightly | 42 | 38
  DAQ, Very slightly | 40 | 39
  IAQ, Slightly | 11 | 28
  DAQ, Slightly | 10 | 24
  IAQ, Neither slightly nor moderately | 2 | 1
  DAQ, Neither slightly nor moderately | 1 | 1
  IAQ, Moderately | 5 | 11
  DAQ, Moderately | 7 | 4
  IAQ, Markedly | 0 | 4
  DAQ, Markedly | 0 | 4
  IAQ, Very markedly | 0 | 1
  DAQ, Very markedly | 0 | 3
Statistical Analysis 1: Comparison: FF 110 µg vs FP 200 µg; Comparison of FF 110 µg and FP 200 µg in IAQ; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; Median Difference (Net) = 0.0
Statistical Analysis 2: Comparison: FF 110 µg vs FP 200 µg; Comparison of FF 110 µg and FP 200 µg in DAQ; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; Median Difference (Net) = 0.0

13. Secondary Outcome: Number of Participants Reported Product Feel Soothing in IAQ and DAQ
Description: Participant response for soothing feel at the end of crossover dosing with FF 110 µg and FP 200 µg was evaluated using IAQ and DAQ having question: Did product feel soothing?. Participants specified their responses on a 6-point scale: 0: none; 1: very slightly; 2: slightly; 3: neither slightly nor moderately; 4: moderately; 5; markedly; 6: very markedly.
Time Frame: Day 1
Population: Per Protocol population comprised of all participants who complete both treatment periods. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | FF 110 µg | FP 200 µg
Number analyzed (Participants) | 121 | 121
Participants
  IAQ, None | 28 | 24
  DAQ, None: number analyzed (Participants) | 120 | 121
  DAQ, None | 26 | 25
  IAQ, Very slight | 28 | 31
  DAQ, Very slight: number analyzed (Participants) | 120 | 121
  DAQ, Very slight | 34 | 31
  IAQ, Slight | 25 | 27
  DAQ, Slight: number analyzed (Participants) | 120 | 121
  DAQ, Slight | 25 | 29
  IAQ, Neither slight nor moderate | 17 | 16
  DAQ, Neither slight nor moderate: number analyzed (Participants) | 120 | 121
  DAQ, Neither slight nor moderate | 15 | 11
  IAQ, Moderate | 15 | 16
  DAQ, Moderate: number analyzed (Participants) | 120 | 121
  DAQ, Moderate | 11 | 19
  IAQ, Marked | 4 | 5
  DAQ, Marked: number analyzed (Participants) | 120 | 121
  DAQ, Marked | 5 | 6
  IAQ, Very marked | 4 | 2
  DAQ, Very marked: number analyzed (Participants) | 120 | 121
  DAQ, Very marked | 4 | 0
Statistical Analysis 1: Comparison: FF 110 µg vs FP 200 µg; This analysis is for IAQ; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.968, Cochran-Mantel-Haenszel; Median Difference (Net) = 0.0
Statistical Analysis 2: Comparison: FF 110 µg vs FP 200 µg; This analysis is for DAQ; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.797, Cochran-Mantel-Haenszel; Mean Difference (Net) = 0.0

14. Secondary Outcome: Number of Participants Reported Product Make Want to Sneeze in IAQ
Description: Participant response regarding sneezing effect at the end of crossover dosing with FF 110 µg and FP 200 µg was evaluated using IAQ having question: Did product make want to sneeze?. Participants specified their responses on a 6-point scale: 0: No urgency; 1: Very slight urgency; 2: slight urgency; 3: Neither slight nor moderate urgency; 4: Moderate urgency; 5; Marked urgency; 6: Very marked urgency.
Time Frame: Day 1
Population: Per protocol population. Only those participants available at the indicated time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | FF 110 µg | FP 200 µg
Number analyzed (Participants) | 121 | 121
Participants
  No urgency | 87 | 93
  Very slight urgency | 17 | 12
  Slight urgency | 8 | 10
  Neither slight nor moderate urgency | 2 | 2
  Moderate urgency | 2 | 2
  Marked urgency | 3 | 2
  Very marked urgency | 2 | 0
Statistical Analysis 1: Comparison: FF 110 µg vs FP 200 µg; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.221, Cochran-Mantel-Haenszel; Median Difference (Net) = 0.0

15. Secondary Outcome: Number of Participants Satisfied With Product in DAQ
Description: Number of participants responding to product satisfaction with delayed attributes questionnaire, Question: How satisfied with product?. Participants specified their responses on a 6-point scale: 0: very satisfied; 1: moderately satisfied; 2: somewhat satisfied; 3: neither satisfied nor dissatisfied; 4: somewhat dissatisfied; 5; moderately dissatisfied; 6: very dissatisfied.
Time Frame: Day 1
Population: Per protocol population. Only those participants available at the indicated time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | FF 110 µg | FP 200 µg
Number analyzed (Participants) | 121 | 120
Participants
  Very satisfied | 44 | 34
  Moderately satisfied | 27 | 23
  Somewhat satisfied | 17 | 27
  Neither satisfied nor dissatisfied | 19 | 21
  Somewhat dissatisfied | 7 | 8
  Moderately dissatisfied | 5 | 7
  Very dissatisfied | 2 | 0
Statistical Analysis 1: Comparison: FF 110 µg vs FP 200 µg; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.205, Cochran-Mantel-Haenszel; Median Difference (Net) = 0.0

16. Secondary Outcome: Number of Participants Reported Nasal Irritation in DAQ
Description: Participant response regarding nasal irritation at the end of crossover dosing with FF 110 µg and FP 200 µg was evaluated using DAQ having question: Did product cause nasal irritation?. Participants specified their responses on a 6-point scale: 0: none; 1: very slight; 2: slight; 3: neither slight nor moderate; 4: moderate; 5; marked; 6: very marked.
Time Frame: Day 1
Population: Per protocol population. Only those participants available at the indicated time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | FF 110 µg | FP 200 µg
Number analyzed (Participants) | 121 | 121
Participants
  None | 89 | 78
  Very slight | 18 | 21
  Slight | 6 | 10
  Neither slight nor moderate | 2 | 3
  Moderate | 3 | 7
  Marked | 2 | 1
  Very marked | 1 | 1
Statistical Analysis 1: Comparison: FF 110 µg vs FP 200 µg; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.108, Cochran-Mantel-Haenszel; Median Difference (Net) = 0.0

17. Secondary Outcome: Number of Participants Reported Nasal Irritation Bothersome in DAQ
Description: Participant response regarding bothersome of nasal irritation at the end of crossover dosing with FF 110 µg and FP 200 µg was evaluated using DAQ having question: How bothersome was nasal irritation?. Participants specified their responses on a 6-point scale: 0: none; 1: very slightly; 2: slightly; 3: neither slightly nor moderately; 4: moderately; 5; markedly; 6: very markedly.
Time Frame: Day 1
Population: Per protocol population. Only those participants available at the indicated time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | FF 110 µg | FP 200 µg
Number analyzed (Participants) | 38 | 48
Participants
  None | 7 | 7
  Very slightly | 15 | 22
  Slightly | 9 | 8
  Neither slightly nor moderately | 2 | 2
  Moderately | 4 | 6
  Markedly | 0 | 1
  Very markedly | 1 | 2
Statistical Analysis 1: Comparison: FF 110 µg vs FP 200 µg; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.694, Cochran-Mantel-Haenszel; Median Difference (Net) = 0.0

18. Secondary Outcome: Number of Participants Comply With Product if Prescribed in DAQ
Description: Number of participants responding to product attributes using delayed attributes questionnaire, Question: How likely to comply if prescribed?. Participants specified their responses on a 6-point scale: 0: very likely; 1: moderately likely; 2: somewhat likely; 3: neither likely nor unlikely; 4: somewhat unlikely; 5; moderately unlikely; 6: very unlikely.
Time Frame: Day 1
Population: Per protocol population. Only those participants available at the indicated time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | FF 110 µg | FP 200 µg
Number analyzed (Participants) | 121 | 120
Participants
  Very likely | 63 | 45
  Moderately likely | 19 | 26
  Somewhat likely | 18 | 16
  Neither likely nor unlikely | 7 | 10
  Slightly unlikely | 4 | 12
  Moderately unlikely | 4 | 7
  Very unlikely | 6 | 4
Statistical Analysis 1: Comparison: FF 110 µg vs FP 200 µg; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.020, Cochran-Mantel-Haenszel; Median Difference (Net) = 0.0

ADVERSE EVENTS:
Time Frame: Adverse events were reported throughout the treatment period (Day 1), as this is single day study which included pre treatment, washout, treatment periods 1 and 2
Description: Intent-to-treat population was used which comprised of all participants who were randomized to study drug, formed the basis for all summaries of safety, background, and demographic data.
Arm/Group | FF 110 µg | FP 200 µg
All-Cause Mortality (participants affected / at risk) | 0/127 | 0/127
Serious Adverse Events (participants affected / at risk) | 0/127 | 0/127
Other Adverse Events (participants affected / at risk) | 3/127 | 0/127
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FF 110 µg (N=127) | FP 200 µg (N=127)
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.